CLINICAL TRIAL: NCT01920048
Title: REVascularisation for Ischaemic VEntricular Dysfunction (REVIVED): a Randomized Comparison of Percutaneous Coronary Intervention (With Optimal Medical Therapy) Versus Optimal Medical Therapy Alone for Treatment of Heart Failure Secondary to Coronary Disease
Brief Title: Study of Efficacy and Safety of Percutaneous Coronary Intervention to Improve Survival in Heart Failure
Acronym: REVIVED-BCIS2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King's College London (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government); London School of Hygiene and Tropical Medicine (Other); University of York (Other); Guy's and St Thomas' NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Divaka Perera, Consultant Cardiologist and Professor of Cardiology, King's College London
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ISRCTN45979711; ISRCTN45979711 (Other: International Standard Randomised Controlled Trial Number Register)
Record Dates: First submitted 2013-08-03; First posted 2013-08-09 (Estimated); Last update posted 2022-05-31 (Actual); Status verified 2022-05

CONDITIONS: Ischemic Cardiomyopathy
Keywords: Heart Failure; Ventricular Dysfunction; Ischemic Cardiomyopathy; Ischemic Heart Disease; Revascularization; Percutaneous Coronary Intervention; Randomized Control Trial; Implantable Cardioverter Defibrillator
MeSH Terms: conditions — Heart Failure; Ventricular Dysfunction; Myocardial Ischemia | interventions — Percutaneous Coronary Intervention; Angioplasty, Balloon; Stents; Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Percutaneous Coronary Intervention and Optimal Medical Therapy (Experimental)
  Interventions: Procedure: Percutaneous Coronary Intervention; Drug: Drug Therapy for Heart Failure; Device: Device Therapy for Heart Failure
- Optimal Medical Therapy alone (Active Comparator)
  Interventions: Drug: Drug Therapy for Heart Failure; Device: Device Therapy for Heart Failure

INTERVENTIONS:
Procedure: Percutaneous Coronary Intervention
  Other Names: Coronary angioplasty/stents
  Arms: Percutaneous Coronary Intervention and Optimal Medical Therapy
Drug: Drug Therapy for Heart Failure — The optimal combination of drugs and doses for each patient will be individualized and will be determined by his/her physician, in accordance with local and international clinical practice guidelines
Device: Device Therapy for Heart Failure — The optimal device therapy for each patient will be individualized and will be determined by his/her physician, in accordance with local and international clinical practice guidelines. In most cases the device will be an Implantable Cardioverter Defibrillator and/or Cardiac Resynchronization Therapy.

SUMMARY:
This study will assess whether percutaneous coronary intervention (angioplasty of the heart arteries) can improve survival and reduce hospitalization in patients with heart failure due to coronary disease, who have been treated with the best contemporary medical therapy.

ELIGIBILITY:
Inclusion Criteria:

ALL of the following:

1. Poor left ventricular function (EF≤35%)
2. Extensive coronary disease
3. Viability in at least 4 dysfunctional segments that can be revascularised by PCI

Exclusion Criteria:

1. Myocardial infarction < 4 weeks prior to randomisation (clinical definition)
2. Decompensated heart failure requiring inotropic support, invasive or non-invasive ventilation or Intra-aortic Balloon Pump/left ventricular assist device therapy <72 hours prior to randomization
3. Sustained Ventricular Tachycardia/Ventricular Fibrillation or appropriate Implantable Cardioverter Defibrillator discharges <72 hours prior to randomization
4. Valve disease requiring intervention
5. Contraindications to percutaneous coronary intervention
6. Age <18 yrs
7. Estimated Glomerular Filtration Rate < 25 ml/min, unless established on dialysis
8. Women who are pregnant
9. Previously enrolled in REVIVED-BCIS2 or current enrollment in other study that may affect REVIVED-BCIS2 outcome data
10. Life expectancy < 1 yr due to non-cardiac pathology

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 700 (Actual)
Dates: Start 2013-08-28 (Actual); Primary Completion 2020-03-19 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
All-cause death or Hospitalization for Heart Failure | 1 to 103 months (min follow-up duration: 24 months)
  This composite endpoint will be collected over the entire duration of follow-up in the trial when the last patient randomized has reached 2 years of follow-up post randomization

SECONDARY OUTCOMES:
Left Ventricular Ejection Fraction | 6 months, 1 year
  Left Ventricular Ejection Fraction (LVEF) on echocardiography
Quality of Life Scores | 6 months, 1 year, 2 years, 3 years, 4 years, 5 years, 6 years, 7 years, 8 years
  Kansas City Cardiomyopathy questionnaire (KCCQ) up to 2 years EuroQol EQ-5D-5L at 6 months and then yearly to the end of follow-up.
New York Heart Association Functional (NYHA) Class | 6 months, 1 year, 2 years
Cardiovascular Death | 1 to 103 months (min follow-up duration: 24 months)
  Cardiovascular death over the entire duration of follow-up
All-cause death | 1 to 103 months (min follow-up duration: 24 months)
  All-cause death over the entire duration of follow-up
Hospitalization due to heart failure | 1 to 103 months (min follow-up duration: 24 months)
  Hospitalization due to heart failure over the entire duration of follow-up
Acute Myocardial Infarction | 1 to 103 months (min follow-up duration: 24 months)
  Acute myocardial infarction (MI) over the entire duration of follow-up
Appropriate Implantable Cardioverter Defibrillator Therapy | 6 months, 1 year, 2 years
  Appropriate implantable cardioverter defibrillator (ICD) therapy to 2 years
Unplanned further revascularization | 1 to 103 months (min follow-up duration: 24 months)
  Unplanned further revascularization over the entire duration of follow-up
Canadian Cardiovascular Society class | 6 months, 1 year, 2 years
  Canadian Cardiovascular Society (CCS) class up to 2 years
Brain-type Natriuretic Peptide level | 6 months, 1 year, 2 years
  Brain natriuretic peptide (BNP or NT-Pro BNP) up to 2 years
Major Bleeding | 6 months, 1 year, 2 years
  Major bleeding up to 2 years

OTHER OUTCOMES:
NHS Resource Use | 1 to 103 months (min follow-up duration: 24 months)
  Health Economic Analysis

CONTACTS AND LOCATIONS:
Overall Officials: Divaka Perera, MB BChir, MA, MD, FRCP, Principal Investigator — King's College London
Locations (40):
- United Kingdom (40):
  - Basingstoke and North Hampshire Hospital, Basingstoke
  - Royal Victoria Hospital, Belfast
  - Birmingham Heartlands Hospital, Birmingham
  - Blackpool Victoria Hospital, Blackpool
  - North Wales Cardiac Centre, Bodelwyddan
  - Royal Bournemouth Hospital, Bournemouth
  - Bristol Heart Institute, Bristol
  - University Hospital Coventry, Coventry
  - Dorset County Hospital, Dorchester
  - Ninewells Hospital, Dundee
  - Royal Infirmary of Edinburgh, Edinburgh
  - Royal Devon and Exeter Hospital, Exeter
  - Golden Jubilee National Hospital, Glasgow
  - Kettering General Hospital, Kettering
  - Leeds General Infirmary, Leeds
  - Glenfield Hospital, Leicester
  - Liverpool Heart and Chest Hospital, Liverpool
  - Barts Heart Centre, London
  - Royal Free Hospital, London
  - Guy's and St Thomas' Hospital, London
  - King's College Hospital, London
  - St George's Hospital, London
  - Manchester Royal Infirmary, Manchester
  - The James Cook University Hospital, Middlesbrough
  - Freeman Hospital, Newcastle
  - Royal Oldham Hospital, Oldham
  - Derriford Hospital, Plymouth
  - Queen Alexandra Hospital, Portsmouth
  - Salisbury District Hospital, Salisbury
  - Northern General Hospital, Sheffield
  - Southampton General Hospital, Southampton
  - Lister Hospital, Stevenage
  - Sunderland Royal Hospital, Sunderland
  - Great Western Hospital, Swindon
  - Pinderfields Hospital, Wakefield
  - New Cross Hospital, Wolverhampton
  - Worcestershire Royal Hospital, Worcester
  - Worthing Hospital, Worthing
  - Wythenshawe Hospital, Wythenshawe
  - York Hospital, York

REFERENCES:
- [Derived] Ovesen C, Dodd M, Ryan M, Clayton T, Sharples L, Perera D. Impact of baseline risk of death or hospitalization on effectiveness of revascularization in patients with ischaemic left ventricular dysfunction-a prespecified analysis of REVIVED-BCIS2. Eur Heart J Qual Care Clin Outcomes. 2025 Dec 19;11(8):1440-1447. doi: 10.1093/ehjqcco/qcaf108. PMID 40972554
- [Derived] Ezad SM, McEntegart M, Dodd M, Didagelos M, Sidik N, Li Kam Wa M, Morgan HP, Pavlidis A, Weerackody R, Walsh SJ, Spratt JC, Strange J, Ludman P, Chiribiri A, Clayton T, Petrie MC, O'Kane P, Perera D; REVIVED-BCIS2 Investigators. Impact of Anatomical and Viability-Guided Completeness of Revascularization on Clinical Outcomes in Ischemic Cardiomyopathy. J Am Coll Cardiol. 2024 Jul 23;84(4):340-350. doi: 10.1016/j.jacc.2024.04.043. Epub 2024 May 15. PMID 38759904
- [Derived] Ryan M, Taylor D, Dodd M, Spertus JA, Kosiborod MN, Shaukat A, Docherty KF, Clayton T, Perera D, Petrie MC; REVIVED-BCIS2 Investigators. Effect of PCI on Health Status in Ischemic Left Ventricular Dysfunction: Insights From REVIVED-BCIS2. JACC Heart Fail. 2024 Sep;12(9):1553-1562. doi: 10.1016/j.jchf.2024.03.010. Epub 2024 Apr 8. PMID 38727649
- [Derived] Chivardi C, Morgan H, Sculpher MJ, Clayton T, Evans R, Dodd M, Petrie M, Rinaldi CA, O'Kane P, Brown L, Perera D, Saramago P; REVIVED-BCIS2 Investigators. Percutaneous Revascularization for Ischemic Left Ventricular Dysfunction: Cost-Effectiveness Analysis of the REVIVED-BCIS2 Trial. Circ Cardiovasc Qual Outcomes. 2024 Jan;17(1):e010533. doi: 10.1161/CIRCOUTCOMES.123.010533. Epub 2023 Nov 6. PMID 37929587
- [Derived] Perera D, Ryan M, Morgan HP, Greenwood JP, Petrie MC, Dodd M, Weerackody R, O'Kane PD, Masci PG, Nazir MS, Papachristidis A, Chahal N, Khattar R, Ezad SM, Kapetanakis S, Dixon LJ, De Silva K, McDiarmid AK, Marber MS, McDonagh T, McCann GP, Clayton TC, Senior R, Chiribiri A; REVIVED-BCIS2 Investigators. Viability and Outcomes With Revascularization or Medical Therapy in Ischemic Ventricular Dysfunction: A Prespecified Secondary Analysis of the REVIVED-BCIS2 Trial. JAMA Cardiol. 2023 Dec 1;8(12):1154-1161. doi: 10.1001/jamacardio.2023.3803. PMID 37878295
- [Derived] Perera D, Morgan HP, Ryan M, Dodd M, Clayton T, O'Kane PD, Greenwood JP, Walsh SJ, Weerackody R, McDiarmid A, Amin-Youssef G, Strange J, Modi B, Lockie T, Hogrefe K, Ahmed FZ, Behan M, Jenkins N, Abdelaal E, Anderson M, Watkins S, Evans R, Rinaldi CA, Petrie MC; REVIVED-BCIS2 Investigators. Arrhythmia and Death Following Percutaneous Revascularization in Ischemic Left Ventricular Dysfunction: Prespecified Analyses From the REVIVED-BCIS2 Trial. Circulation. 2023 Sep 12;148(11):862-871. doi: 10.1161/CIRCULATIONAHA.123.065300. Epub 2023 Aug 9. PMID 37555345
- [Derived] Ezad SM, Ryan M, Perera D. Can Percutaneous Coronary Intervention Revive a Failing Heart? Heart Int. 2022 Dec 21;16(2):72-74. doi: 10.17925/HI.2022.16.2.72. eCollection 2022. PMID 36741102
- [Derived] Perera D, Clayton T, O'Kane PD, Greenwood JP, Weerackody R, Ryan M, Morgan HP, Dodd M, Evans R, Canter R, Arnold S, Dixon LJ, Edwards RJ, De Silva K, Spratt JC, Conway D, Cotton J, McEntegart M, Chiribiri A, Saramago P, Gershlick A, Shah AM, Clark AL, Petrie MC; REVIVED-BCIS2 Investigators. Percutaneous Revascularization for Ischemic Left Ventricular Dysfunction. N Engl J Med. 2022 Oct 13;387(15):1351-1360. doi: 10.1056/NEJMoa2206606. Epub 2022 Aug 27. PMID 36027563
- [Derived] Perera D, Clayton T, Petrie MC, Greenwood JP, O'Kane PD, Evans R, Sculpher M, Mcdonagh T, Gershlick A, de Belder M, Redwood S, Carr-White G, Marber M; REVIVED investigators. Percutaneous Revascularization for Ischemic Ventricular Dysfunction: Rationale and Design of the REVIVED-BCIS2 Trial: Percutaneous Coronary Intervention for Ischemic Cardiomyopathy. JACC Heart Fail. 2018 Jun;6(6):517-526. doi: 10.1016/j.jchf.2018.01.024. PMID 29852933